CLINICAL TRIAL: NCT06913972
Title: A Comparative Analysis of Myopia Prevalence Among Madarsa Students vs. Non-Madarsa Students in Sukkur
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSRSW/Batch-Fall23/812
Record Dates: First submitted 2025-03-29; First posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myopia (nearsightedness) has become a major global health concern, particularly among students, due to factors such as prolonged screen time, close-up work, and limited outdoor activities. In regions like Sukkur, Pakistan, the educational environments and lifestyles of students in Madarsas (religious schools) differ significantly from those in non-Madarsa (regular) schools, potentially influencing the prevalence of myopia. This comparative cross-sectional study aims to assess and compare the prevalence of myopia among Madarsa and non-Madarsa students in Sukkur.

DETAILED DESCRIPTION:
The study will be conducted at Al Shifa Trust Eye Hospital over six months, involving students aged 5-20 years. Informed consent will be obtained from parents or guardians, and a structured questionnaire will collect data on lifestyle factors such as time spent on near work, outdoor activities, family history of refractive errors, and the use of corrective eyewear. Visual acuity and refractive errors will be assessed using standard eye charts, cycloplegic refraction, and measurements of keratometry, biometry, and axial length. The data will be analyzed using descriptive statistics, including frequencies, means, and standard deviations, with normality tests applied to continuous variables. Chi-square tests and Independent t-tests will be used for comparative analysis, while logistic regression will assess risk factors associated with myopia. The study will help determine the prevalence of myopia and its contributing factors in these student populations, informing potential interventions.

ELIGIBILITY:
Inclusion Criteria:

* Students aged 5-20 years.[18]
* Students of Sukkur enrolled in either Madarsa or schools.
* Parents or guardians who understand and sign the informed consent form.
* Students who are willing to undergo an eye examination and complete the research

Exclusion Criteria:

* Students with known systemic diseases or eye conditions (e.g., cataracts, retinal diseases) that could influence the assessment of myopia.
* Students who have had corrective eye surgery (e.g., LASIK) or those who have worn contact lenses or glasses for less than 3 months.
* Students unable to participate due to language barriers or other communincation difficulties
* Students with neurological conditions affecting vision
* Students unable to cooperate with visual acuity testing due to cognitive impairments"

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: To compare the prevalence of myopia among Madarsaand schoolstudents in Sukkur.
Sampling Method: Non-Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
refraction | 12 Months
  In the eye, refraction is the bending of light rays as they pass through the cornea and lens, focusing them onto the retina for clear vision
auto-refractometer | 12 Months
  An auto-refractometer is a device used in eye exams to objectively measure a person's refractive error and determine the prescription needed for glasses or contact lenses, by analyzing how light reflects off the eye

CONTACTS AND LOCATIONS:
Locations (1):
- Al Shifa trust eye Hospital, Sukkur, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No